CLINICAL TRIAL: NCT04720131
Title: Camrelizumab Combined With Apatinib and Capecitabine for Patients With Advanced Biliary Tract Cancer: a Phase 2, Single-arm, Prospective Study.
Brief Title: Camrelizumab Combined With Apatinib and Capecitabine in Patients With Advanced Biliary Tract Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-BTC＆PD-1
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Biliary Tract Cancer; Anti-PD-1 Therapy; Targeted Molecular Therapy; Capecitabine
Keywords: Capecitabine; Targeted Molecular Therapy; Biliary Tract Cancer; Camrelizumab
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — camrelizumab; apatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab combined with Apatinib and Capecitabine (Experimental): Camrelizumab was administered 200mg iv every 3 weeks. Capecitabine was administered 1000mg/m2 orally, b.i.d. every 3 weeks (Day 1-14 of a treatment cycle) Apatinib:A safety-run-in was conducted in the first cycle to identify the recommended dose of Apatinib, the initial dose was administered 250mg orally daily every 3 weeks (Day 1-14 of a treatment cycle). The dose of Apatinib increase and reduction was 250 mg orally q.d. and 250 mg orally q.o.d. every 3 weeks respectively according to the number of doses limiting toxicity events (DLTs) in the initial group. The final dose of Apatinib for the extension stage was detemained by the result of safety-run-in stage.
  Interventions: Drug: Camrelizumab; Drug: apatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab was administered 200mg iv every 3 weeks.
Drug: apatinib — Apatinib A safety-run-in was conducted in the first cycle to identify the recommended dose of Apatinib, the initial dose was administered 250mg orally daily every 3 weeks (Day 1-14 of a treatment cycle) The dose of Apatinib increase and reduction was 250 mg orally q.d. and 250 mg orally q.o.d. every 3 weeks respectively according to the number of doses limiting toxicity events (DLTs) in the initial group.
  The final dose of Apatinib for the extension stage was detemained by the result of safety-run-in stage.
Drug: Capecitabine — Capecitabine was administered 1000mg/m2 orally, b.i.d. every 3 weeks (Day 1-14 of a treatment cycle)

SUMMARY:
Biliary tract cancer (BTC) is a series of rare malignancies with poor overall prognosis. Radical surgery the preferred treatment option, but most patients have lost the opportunity of surgery at the time of diagnosis. At present, there are limited systematical treatment options for biliary tract cancer, with poor efficacy and short duration of responses. In the past few years, immune checkpoint inhibitors (ICIs) therapy has gradually been added to the advanced biliary comprehensive treatment. However, in view of the low incidence and high heterogeneity of BTC, more large number of clinical trials and practices need to be carried out, and the effective combination regimens and predictive biomarkers need to be explored. This study is a single-arm, open-label, prospective cohort study, combining Camrelizumab with apatinib and capecitabine as the first-line or second-line treatment for patients with advanced biliary tract cancer. The study aims to explore the efficacy and safety of the combination regimen, and try to find biomarkers that can guild treatment. In this study, 34 patients were enrolled by the Simon's two-stage design, with the objective response rate as the primary endpoint and the disease control rate, progression-free survival, overall survival and safety as secondary endpoints. It is expected that the three-drug combination regimen will have significant efficacy and manageable adverse reactions, and predictive biomarkers can be found.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old, both genders.
* Conform to the histological or cytological confirmation of biliary tract carcinoma，including gallbladder cancers and cholangiocarcinomas.
* Patients have advanced unresectable biliary tract carcinoma, including recurrence or metastasis of BTC after radical resection.
* Patientss who have not received any prior PD-1 inhibitor and Apatinib therapy.
* Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1within one week before enrollment.
* Life expectancy greater than 3 months.
* Patient must have adequate organ function defined by the study-specified laboratory tests.
* Patient must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or planned transplantation.
* Patients with other malignant tumor in the past 5 years (except cured skin basal cell carcinoma and cervical carcinoma).
* History of esophageal variceal bleeding, hepatic encephalopathy, massive ascites and abdominal infection.
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 14 days before study drug administration.
* Known history of hypersensitivity to any components of the camrelizumab, apatinib and Capecitabine formulation, or other antibody formulation.
* Patients who may receive live vaccine during the study, or previous had vaccination within 4 weeks.
* Known or occurrence of central nervous system (CNS) metastases or hepatic encephalopathy.
* Peripheral neuropathy> Grade 1.
* Patients with any active autoimmune disease or history of autoimmune disease.
* History of immunodeficiency or human immunodeficiency virus (HIV) infection.
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention.
* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
* Coagulation abnormalities (INR>1.5 or APTT>1.5×ULN), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
* History of hereditary or acquired bleeding and thrombotic tendency, such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.
* Patients with obvious cough blood or hemoptysis volume of half teaspoon (2.5 ml) or more within 2 months before entering the study.
* Have significant clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before entering the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood++ and above at baseline, or vasculitis, etc.
* Previous Arterial/venous thrombosis events within 6 months.
* Required for long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).
* Severe infection within 4 weeks before the first medication (e.g. need for intravenous antibiotics, antifungal or antiviral drugs), or active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing.
* Participated in any other drug clinical study within 4 weeks before the first administration, or no more than 5 half lives from the last administration.
* Known history of psychotropic drug abuse or drug abuse.
* Pregnant and lactating women. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 30 months
  The proportion of patients with measurable disease who achieved complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Disease Control Rates (DCR) | 30 months
  The proportion of patients achieving CR or PR or stable disease (SD)
Progression-Free Survival | 30 months
  The duration from the beginning of the treatment to the disease progression, or death from any cause, or last progression-free survival assessment for patients alive without progression
Overall Survival | 30 months
  The duration from the enrollment to death from any cause
Safety | 30 months
  The incidence of any grade treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Deng, Principal Investigator — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be obtained with the consent of the principal investigator

REFERENCES:
- [Background] de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999 Oct 28;341(18):1368-78. doi: 10.1056/NEJM199910283411807. No abstract available. PMID 10536130
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Razumilava N, Gores GJ. Cholangiocarcinoma. Lancet. 2014 Jun 21;383(9935):2168-79. doi: 10.1016/S0140-6736(13)61903-0. Epub 2014 Feb 26. PMID 24581682
- [Background] Ilyas SI, Khan SA, Hallemeier CL, Kelley RK, Gores GJ. Cholangiocarcinoma - evolving concepts and therapeutic strategies. Nat Rev Clin Oncol. 2018 Feb;15(2):95-111. doi: 10.1038/nrclinonc.2017.157. Epub 2017 Oct 10. PMID 28994423
- [Background] Everhart JE, Ruhl CE. Burden of digestive diseases in the United States Part III: Liver, biliary tract, and pancreas. Gastroenterology. 2009 Apr;136(4):1134-44. doi: 10.1053/j.gastro.2009.02.038. Epub 2009 Feb 24. No abstract available. PMID 19245868
- [Background] Jusakul A, Cutcutache I, Yong CH, Lim JQ, Huang MN, Padmanabhan N, Nellore V, Kongpetch S, Ng AWT, Ng LM, Choo SP, Myint SS, Thanan R, Nagarajan S, Lim WK, Ng CCY, Boot A, Liu M, Ong CK, Rajasegaran V, Lie S, Lim AST, Lim TH, Tan J, Loh JL, McPherson JR, Khuntikeo N, Bhudhisawasdi V, Yongvanit P, Wongkham S, Totoki Y, Nakamura H, Arai Y, Yamasaki S, Chow PK, Chung AYF, Ooi LLPJ, Lim KH, Dima S, Duda DG, Popescu I, Broet P, Hsieh SY, Yu MC, Scarpa A, Lai J, Luo DX, Carvalho AL, Vettore AL, Rhee H, Park YN, Alexandrov LB, Gordan R, Rozen SG, Shibata T, Pairojkul C, Teh BT, Tan P. Whole-Genome and Epigenomic Landscapes of Etiologically Distinct Subtypes of Cholangiocarcinoma. Cancer Discov. 2017 Oct;7(10):1116-1135. doi: 10.1158/2159-8290.CD-17-0368. Epub 2017 Jun 30. PMID 28667006
- [Background] Weinberg BA, Xiu J, Lindberg MR, Shields AF, Hwang JJ, Poorman K, Salem ME, Pishvaian MJ, Holcombe RF, Marshall JL, Morse MA. Molecular profiling of biliary cancers reveals distinct molecular alterations and potential therapeutic targets. J Gastrointest Oncol. 2019 Aug;10(4):652-662. doi: 10.21037/jgo.2018.08.18. PMID 31392046
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Kim R, Coppola D, Wang E, Chang YD, Kim Y, Anaya D, Kim DW. Prognostic value of CD8CD45RO tumor infiltrating lymphocytes in patients with extrahepatic cholangiocarcinoma. Oncotarget. 2018 May 4;9(34):23366-23372. doi: 10.18632/oncotarget.25163. eCollection 2018 May 4. PMID 29805739
- [Background] Chen X, Wu X, Wu H, Gu Y, Shao Y, Shao Q, Zhu F, Li X, Qian X, Hu J, Zhao F, Mao W, Sun J, Wang J, Han G, Li C, Xia Y, Seesaha PK, Zhu D, Li H, Zhang J, Wang G, Wang X, Li X, Shu Y. Camrelizumab plus gemcitabine and oxaliplatin (GEMOX) in patients with advanced biliary tract cancer: a single-arm, open-label, phase II trial. J Immunother Cancer. 2020 Nov;8(2):e001240. doi: 10.1136/jitc-2020-001240. PMID 33172881
- [Background] Piha-Paul SA, Oh DY, Ueno M, Malka D, Chung HC, Nagrial A, Kelley RK, Ros W, Italiano A, Nakagawa K, Rugo HS, de Braud F, Varga AI, Hansen A, Wang H, Krishnan S, Norwood KG, Doi T. Efficacy and safety of pembrolizumab for the treatment of advanced biliary cancer: Results from the KEYNOTE-158 and KEYNOTE-028 studies. Int J Cancer. 2020 Oct 15;147(8):2190-2198. doi: 10.1002/ijc.33013. Epub 2020 May 2. PMID 32359091
- [Background] Manegold C, Dingemans AC, Gray JE, Nakagawa K, Nicolson M, Peters S, Reck M, Wu YL, Brustugun OT, Crino L, Felip E, Fennell D, Garrido P, Huber RM, Marabelle A, Moniuszko M, Mornex F, Novello S, Papotti M, Perol M, Smit EF, Syrigos K, van Meerbeeck JP, van Zandwijk N, Yang JC, Zhou C, Vokes E. The Potential of Combined Immunotherapy and Antiangiogenesis for the Synergistic Treatment of Advanced NSCLC. J Thorac Oncol. 2017 Feb;12(2):194-207. doi: 10.1016/j.jtho.2016.10.003. Epub 2016 Oct 8. PMID 27729297
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Kim ST, Kang JH, Lee J, Lee HW, Oh SY, Jang JS, Lee MA, Sohn BS, Yoon SY, Choi HJ, Hong JH, Kim MJ, Kim S, Park YS, Park JO, Lim HY. Capecitabine plus oxaliplatin versus gemcitabine plus oxaliplatin as first-line therapy for advanced biliary tract cancers: a multicenter, open-label, randomized, phase III, noninferiority trial. Ann Oncol. 2019 May 1;30(5):788-795. doi: 10.1093/annonc/mdz058. PMID 30785198
- [Background] Kim RD, Chung V, Alese OB, El-Rayes BF, Li D, Al-Toubah TE, Schell MJ, Zhou JM, Mahipal A, Kim BH, Kim DW. A Phase 2 Multi-institutional Study of Nivolumab for Patients With Advanced Refractory Biliary Tract Cancer. JAMA Oncol. 2020 Jun 1;6(6):888-894. doi: 10.1001/jamaoncol.2020.0930. PMID 32352498
- [Background] Lin J, Yang X, Long J, Zhao S, Mao J, Wang D, Bai Y, Bian J, Zhang L, Yang X, Wang A, Xie F, Shi W, Yang H, Pan J, Hu K, Guan M, Zhao L, Huo L, Mao Y, Sang X, Wang K, Zhao H. Pembrolizumab combined with lenvatinib as non-first-line therapy in patients with refractory biliary tract carcinoma. Hepatobiliary Surg Nutr. 2020 Aug;9(4):414-424. doi: 10.21037/hbsn-20-338. PMID 32832493
- [Derived] Jing C, Bai Z, Tong K, Yang X, Liu K, Wu H, Zhu J, Guo W, Zhang Z, Deng W. Efficacy and safety of camrelizumab, apatinib, and capecitabine combination therapy in advanced biliary tract cancer: a phase 2, nonrandomized, prospective study. Oncologist. 2024 Nov 4;29(11):e1565-e1574. doi: 10.1093/oncolo/oyae154. PMID 39102756